CLINICAL TRIAL: NCT03128658
Title: Trauma Induced Coagulopathy and Inflammation
Acronym: TrICI
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Collaborators: Princeton University (Other)
Responsible Party: Sponsor
Other Study IDs: 826515
Record Dates: First submitted 2017-03-15; First posted 2017-04-25 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2021-03

CONDITIONS: Trauma Injury; Trauma; Coagulopathy
Keywords: Trauma induced coagulopathy
MeSH Terms: conditions — Accidental Injuries; Wounds and Injuries; Hemostatic Disorders | interventions — Thrombelastography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — During the initial trauma evaluation, 15 ml of blood will be collected for research purposes during the routine blood trauma blood draw. Additional 15 ml samples will be collected at 3 hours, 6 hours, 12 hours, 24 hours, 48 hours and 5 days post admission.
  Blood samples will be analyzed for coagulation parameters using thromboelastography.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Trauma patients: Trauma patients with a systolic blood pressure of 90 mmHg or less, in need for blood product transfusion within 1 hour of admission, and/or an ISS (injury severity score) of greater than or equal to 15.
  Interventions: Diagnostic Test: Thromboelastography; Diagnostic Test: Computational model

INTERVENTIONS:
Diagnostic Test: Thromboelastography — Thromboelastography (TEG) tests for parameters related to efficiency of blood coagulation. The parameters are: reaction time (R value), the K value, the angle and the maximum amplitude (MA)
Diagnostic Test: Computational model — The computational whole-patient systems model is a multiscale, multi-compartment model whose state-space is defined by a very large and heterogeneous set of variables as well as a large number of input parameters. The model will be integrated in time for various initial trauma conditions in an attempt to determine whether the model can be predictive, and help us discover new variables that are more predictive of clinical outcomes than those employed in current clinical protocols.

SUMMARY:
While a number of factors are known to be associated with the development of trauma induced coagulopathy (TIC), inflammation, and multi-organ failure, we currently cannot predict which patients are at risk for developing these life threatening conditions with any certainty. In this prospective observational study, we will investigate the many factors that contribute to the development of trauma induced coagulopathy, post injury inflammation and the development of organ dysfunction in order to develop a multi scale computational algorithm of clinical prediction. Using a convenience sample technique, demographic data, physiologic data, blood samples and clinical variables will be collected over 5 days following traumatic injury. A computational model will be used to predict the development of TIC and multi-organ failure.

DETAILED DESCRIPTION:
A prospective, observational, convenience sample of trauma patients 18 years old or older who present to the trauma bay as a trauma alert will be included after evaluation by the on-call trauma surgeon and research assistant. Minimally injured patients will be compared to those with a systolic blood pressure of 90 mmHg or less, the need for blood product transfusion within 1 hour of admission, and/or an ISS (injury severity score) of greater than or equal to 15. Demographic data including past medical/medication history as well as clinical data including continuous vital signs will be recorded. If eligibility criteria are met, the research blood samples will be drawn at the same time as routine clinical samples. Blood samples (approximately 15 ml) will be taken on admission, 3hr, 6hrs, 12hrs, 24 hrs, 48 hrs, and 5 days post admission. Vital signs, number of blood transfusions, volume of crystalloid, administration of medications, and the values of routine laboratories will be monitored continuously for 24 hours, and then cumulatively for up to 5 days. After the last blood draw, we will be following the patient's outcome for up to 30 days. If patients are discharged or die prior to completing the 5 days of blood samples, additional samples and/or clinic appointments for the purpose of research will not be obtained. A computational algorithm will be used to predict the development of trauma induced coagulopathy, inflammation and multi-organ failure.

ELIGIBILITY:
Inclusion Criteria:

* Injured patients presenting to the trauma bay with a trauma alert activation (highest level of activation)
* Age 18 years old or more

Exclusion Criteria:

* Transfer duration to trauma service exceeding 6 hours.
* Known pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Trauma patients 18 years or older who present to the trauma bay as a trauma alert (highest level of activation), requiring blood product transfusion within 1 hour of admission, and/or having an injury severity score (ISS) greater than or equal to 15.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2017-02-27 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Thromboelastography parameters T0 -T3 | Between time of admission (T0) and 3 hours (T3)
  Variables: Reaction time (R value), the K value, the angle and the maximum amplitude (MA)
Change in Thromboelastography parameters T3 -T6 | Between 3 hours (T3) and 6 hours (T6)
  Variables: Reaction time (R value), the K value, the angle and the maximum amplitude (MA)
Change in Thromboelastography parameters T6 -T12 | Between 6 hours (T6) and 12 hours (T12)
  Variables: Reaction time (R value), the K value, the angle and the maximum amplitude (MA)
Change in Thromboelastography parameters T12 - T24 | Between 12 hours (T12) and 24 hours (T24)
  Variables: Reaction time (R value), the K value, the angle and the maximum amplitude (MA)
Change in Thromboelastography parameters T24 - T48 | Between 24 hours (T24) and 48 hours (T48)
  Variables: Reaction time (R value), the K value, the angle and the maximum amplitude (MA)
Change in Thromboelastography parameters T48 - T120 | Between 48 hours (T48) and 120 hours (T120)
  Variables: Reaction time (R value), the K value, the angle and the maximum amplitude (MA)

CONTACTS AND LOCATIONS:
Locations (1):
- Penn Presbyterian Medical Center, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-08-02): https://cdn.clinicaltrials.gov/large-docs/58/NCT03128658/Prot_SAP_000.pdf
  • Informed Consent Form (2018-12-18): https://cdn.clinicaltrials.gov/large-docs/58/NCT03128658/ICF_001.pdf